CLINICAL TRIAL: NCT05630937
Title: Phase I/II Study on Safety and Efficacy of NMS-01940153E in Adult Patients With Unresectable Hepatocellular Carcinoma (HCC) Previously Treated With Systemic Therapy
Brief Title: Study on Safety and Efficacy of NMS-01940153E in Adult Patients With Unresectable Hepatocellular Carcinoma (HCC) Previously Treated With Systemic Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: In the Phase II part of the study, among the participants evaluable for efficacy, no objective (partial response or clinical response) was observed at the first futility analysis.
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MPSA-153-001; 2020-001002-26 (EudraCT Number)
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC)
Keywords: Unresectable Hepatocellular Carcinoma (HCC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMS-01940153E (Experimental): Phase I: Patients will be allocated to sequential cohorts of progressively higher dose levels of NMS-01940153E based on the presence of Dose Limiting Toxicities (DLT).
  Phase II: Patients will be treated at the recommended Phase II dose (RP2D) defined in the Phase I portion.
  Interventions: Drug: NMS-01940153E

INTERVENTIONS:
Drug: NMS-01940153E — Route of administration: intravenous (IV) solution

SUMMARY:
This is a Phase I/II, open-label, non-randomized, multicenter study to explore safety, tolerability and antitumor activity of NMS-01940153E as single agent in adult patients with unresectable hepatocellular carcinoma (HCC) previously treated with systemic therapy.

The Phase I portion is designed as a dose-escalation study in sequential cohorts of patients aimed to obtain the maximum tolerated dose (MTD) that is defined based on the dose limiting toxicities (DLTs) observed in the first cycle of treatment.

The Phase II portion is designed as a two-stage study with an interim analysis for futility and stopping criteria for unacceptable toxicity to assess the antitumor activity of NMS-01940153E in adult patients with unresectable HCC previously treated with systemic therapy measured as objective response rate.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Histological, cytological or radiological diagnosis of HCC, according to the American Association for the Study of Liver Diseases (AASLD) / European Association for the Study of the Liver (EASL) criteria, in subjects that are refractory or not able to tolerate the standard therapy, or subjects for whom the standard therapy is not considered appropriate by the physician.
2. The subject has disease that is not amenable to a curative treatment approach (e.g., transplant, surgery, radiofrequency ablation) and unsuitable for or refractory to locoregional treatments (e.g., TACE).
3. At least one uni-dimensional measurable lesion by CT or MRI according to RECIST 1.1 which is either not previously treated by local therapy or, if treated, it has clearly progressed before the subject is recruited.
4. Phase I only: subjects must have disease relapsed or refractory to the standard of care treatment not exceeding 3 lines of prior systemic treatment. Subjects intolerant to previous treatment with tyrosine kinase inhibitors (TKIs) are eligible. Phase II: subjects must have disease relapsed or refractory to the standard of care treatment including an immunocheckpoint inhibitor as first line and at least a tyrosine kinase inhibitor, not exceeding 3 lines of prior systemic treatment. A minimum of 14 days of treatment with prior TKI would be required to qualify as line of therapy;
5. Child-Pugh score ≤ 6 (class A).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Age ≥18 years old on day of consent.
8. No history of liver transplantation or not listed for high urgent transplantation.
9. Meets required laboratory data
10. In case of active hepatitis B (HBV) or chronic HIV infection the patient should receive antiviral therapy per local standard of care.
11. Patients must use effective contraception or abstinence. Female subjects must be surgically sterile or, if subjects of childbearing potential, must agree to use effective contraception or abstinence during the period of therapy and in the following 180 days after discontinuation of study treatment. Male subjects must be surgically sterile or must agree to use effective contraception or abstinence during the period of therapy and in the following 90 days after discontinuation of study treatment.
12. With the exception of alopecia, resolution of all acute toxic effects of any prior systemic therapy, surgery or radiotherapy to National Cancer Institute (NCI) common terminology criteria (CTC) (Version 5.0) Grade ≤1 or to the baseline laboratory values as defined in Inclusion Criterion Number 9.
13. Able and willing to comply with scheduled visits, therapy plans, and laboratory tests required in this protocol.
14. Signed and dated independent ethics committee (IEC)-approved Informed Consent Form indicating that the subject is aware of the neoplastic nature of his/her disease and has been informed of the procedures to be followed, the investigational nature of the therapy, potential benefits, side effects, discomforts, risks and alternative treatments.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

1. Known fibrolamellar HCC or mixed hepato-cholangiocarcinoma.
2. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding are excluded with the following clarification: subjects with history of prior variceal bleeding must have been treated with adequate endoscopic therapy without any evidence of recurrent bleeding for at least 6 months prior to study entry and must be stable on optimal medical management (e.g. non-selective beta blocker, proton pump inhibitor) at study entry.
3. Subjects with QT interval using Fridericia standard (QTcF) ≥480 milliseconds or with risk factors for torsade de pointes (e.g., heart failure, uncontrolled hypokalemia, family history of long QT syndrome) or receiving treatment with concomitant medications known to prolong the QT/QTc interval that cannot be replaced with another treatment.
4. Ascites defined as CTCAE Grade ≥2. Subjects who have been on a stable medication regimen for at least 2 months to manage ascites are eligible if they show ascites Grade <2.

   Subjects with clinically undetectable ascites who are Child A with detectable ascites at CT/MRI are eligible.
5. Uncontrolled high blood pressure (systolic blood pressure, SBP >150 mmHg and/or diastolic blood pressure, DBP >95 mmHg, despite optimal treatment, on at least 2 out of 3 determinations repeated at 30 minutes interval and done in case that the first one meets the criterion for exclusion).
6. Direct-Acting Antivirals (DAA) at the time of treatment start; previous hepatitis C virus (HCV) treatment with DAAs is allowed.
7. Clinical evidence of hepatic encephalopathy.
8. Known brain metastases or evidence of leptomeningeal disease.
9. Known history of allergic reactions to polysorbate 80.
10. Any of the following in the past 6 months: myocardial infarction, uncontrolled cardiac arrhythmia, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis (except chronic/stable portal vein thrombosis).
11. Major surgery, other than diagnostic surgery, within 4 weeks before treatment start.
12. Any anticancer agent within 4 weeks or, in absence of toxicity, 5 half-lives (within 6 weeks for nitrosureas, mitomycin C and liposomal doxorubicin) before treatment start.
13. Radiation therapy within 4 weeks or radionuclide treatment (e.g., I-131 or Y-90) within 6 weeks before treatment start.
14. Untreated uncontrolled bacterial, viral, or fungal infections including acute HIV infection or acquired immunodeficiency syndrome (AIDS), untreated uncontrolled HBV, untreated uncontrolled HCV, untreated uncontrolled concomitant HBV and HCV; patients who are seropositive following HBV vaccine are eligible.
15. Subjects under treatment with therapeutic dose of anticoagulants (e.g., warfarin or warfarin-related agents, low-molecular weight heparin, or similar agent such as anti Xa and anti-thrombin agents) or antiplatelet agents (e.g. clopidogrel) or with coagulation disorders. Aspirin at dose up to 100 mg is permitted. Prophylaxis with anticoagulants is allowed to meet the international normalized ratio (INR) value range as cited in inclusion criterion 9.
16. Uncontrolled diabetes mellitus.
17. Pregnant or breast-feeding women.
18. Known second malignancy that is progressing or requiring active treatment. Exceptions include adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri.
19. Current enrollment or participation in another interventional clinical trial.
20. Clinically significant respiratory or metabolic diseases uncontrolled by medication.
21. Subjects with active alcohol and/or substances abuse.
22. Any known organ dysfunction, serious illness, acute or chronic medical or psychiatric condition, or laboratory abnormality which, in the Investigator's opinion, may increase the risk associated/interfere with study participation, or with the interpretation of the results.
23. Subjects who, within 7 days prior to the first NMS-01940153E intake, are receiving or received strong inducers of flavin-containing monooxygenase FMO1 and FMO3.
24. Subjects who are receiving sensitive CYP3A4 substrates, CYP3A4 and breast cancer resistance protein (BCRP) substrates with narrow therapeutic index (NTI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - University of California Irvine Health, Orange, California
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
- Italy (6):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Sanitaria Locale Napoli 1 Centro - Ospedale del Mare, Naples
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Pisa
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Participants: 100 mg/m2/Week: All participants in Phase I who received 100 mg/m2/week intravenous NMS-01940153E.
- Phase I Participants: 135 mg/m2/Week: All participants in Phase I who received 135 mg/m2/week intravenous NMS-01940153E.
- Phase II Participants: 100 mg/m2/Week: All participants in Phase II who received 100 mg/m2/week intravenous NMS-01940153E.
- Enrolled But Not Treated: Participants who were enrolled but not randomized and did not receive treatment.
Period: Overall Study
Arm/Group | Phase 1 Participants: 100 mg/m2/Week | Phase I Participants: 135 mg/m2/Week | Phase II Participants: 100 mg/m2/Week | Enrolled But Not Treated
Started | 6 | 6 | 18 | 1
Completed (All participants who completed the study were followed up until death.) | 5 | 5 | 9 | 0
Not Completed | 1 | 1 | 9 | 1
Not completed — Study terminated by sponsor | 1 | 1 | 8 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Enrolled but not treated | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Phase I Participants: 100 mg/m2/Week: All participants in Phase I who received 100 mg/m2/week intravenous NMS-01940153E
- Phase I Treated Participants: 135 mg/m2/Week: All participants in Phase I who received 135 mg/m2/week intravenous NMS-01940153E
- Total: Total of all reporting groups
Arm/Group | Phase I Participants: 100 mg/m2/Week | Phase I Treated Participants: 135 mg/m2/Week | Phase II Participants: 100 mg/m2/Week | Total
Number analyzed (Participants) | 6 | 6 | 18 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 10 | 16
  >=65 years | 3 | 3 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 5 | 6 | 17 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 6 | 18 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Eastern cooperative oncology group performance status [Number; unit: participants] — ECOG PS 0 = Fully active, able to carry on all pre-disease performance without restriction ECOG PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  participants
    ECOG Performance Status 0 | 3 | 3 | 10 | 16
    ECOG Performance Status 1 | 3 | 3 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase I Drug Related Dose Limiting Toxicities (DLTs)
Description: All 12 Phase I treated patients were evaluable for DLT (Dose-Limiting Toxicity Evaluable Set) and included 6 patients treated at each of the two dose levels explored (i.e., 100 mg/m2/week and 135 mg/m2/week) who received at least 66% of the study drug in the first 28-day cycle of treatment and underwent a DLT assessment within the DLT window.
  Participants who experienced DLTs are presented.
Time Frame: Phase I: From screening to end of first 28-day cycle (17 months)
Population: Phase I treated participants
Measure: Count of Participants; unit: Participants
Groups:
- 100 mg/m2/Week Dose (Phase I): All participants in Phase I who received 100 mg/m2/week intravenous NMS-01940153E
- 135 mg/m2/Week Dose (Phase I): All participants in Phase I who received 135 mg/m2/week intravenous NMS-01940153E
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 2

2. Primary Outcome: Phase II Objective Response Rate
Description: The objective response rate (ORR) was calculated as the proportion of evaluable patients who achieved, as best overall response (BOR), confirmed complete response (CR) or partial response (PR) measured by investigator-assessed RECIST 1.1 (Phase II).
Time Frame: Phase II: From Phase II start to Study Completion (23 months)
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Groups:
- Phase II (Evaluable Population): All participants in Phase II who received 100 mg/m2/week intravenous NMS-01940153E in the Evaluable Population.
  The Evaluable Population was participants of the treated set who had measurable disease at baseline assessed according to RECIST 1.1 and at least one tumor evaluation on treatment, unless they died before the first tumor on-treatment assessment, in which case they were considered treatment failure.
Arm/Group | Phase II (Evaluable Population)
Number analyzed (Participants) | 14
Participants
  Stable Disease | 3
  Progressive Disease | 11
  Complete Response | 0
  Partial Response | 0

3. Secondary Outcome: Treatment-emergent Adverse Events by Maximum CTC Grade
Description: The maximum Common Terminology Criteria (CTC) grade (graded using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0) experienced by each participant is presented. If an AE was reported for a participant more than once during treatment, the worst CTC Grade is presented here. Phase 2 started before Phase 1 completed.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: Phase I: From the Study Start Date to Phase I Completion (32 months) - Phase II: From Phase II start to Study Completion (23 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I) | Phase II (Evaluable Population)
Number analyzed (Participants) | 6 | 6 | 18
Participants
  Grade 1 | 0 | 0 | 3
  Grade 2 | 1 | 1 | 8
  Grade 3 | 3 | 3 | 7
  Grade 4 | 1 | 2 | 0

4. Secondary Outcome: Treatment-emergent Adverse Events Related to NMS-01940153E
Description: The number of treatment-emergent adverse events related to NMS-01940153E by maximum CTC grade experienced (graded using NCI CTCAE Version 5.0). Whether the the AE was related or not was assessed by the investigator. If an AE was reported for a participant more than once during treatment, the worst CTC Grade is presented.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening. Phase 2 started before Phase 1 completed.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Number; unit: events
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I) | Phase II (Evaluable Population)
Number analyzed (Participants) | 6 | 6 | 18
events
  Grade 1 | 0 | 0 | 7
  Grade 2 | 1 | 1 | 3
  Grade 3 | 2 | 2 | 2
  Grade 4 | 1 | 2 | 0

5. Secondary Outcome: Hematology: Overall Treatment-emergent Abnormalities by Dose Level and Maximum CTC Grade
Description: Number of treatment emergent abnormalities (at any grade) at all dose levels are presented.
  CTC = Common Terminology Criteria WBC = white blood cells
Time Frame: From screening to 28 days follow-up, an average 6 months
Population: All treated participants
Measure: Number; unit: events
Groups:
- 100 mg/m2/Week Dose (Phase I and II): All participants in Phase I and II who received 100 mg/m2/week intravenous NMS-01940153E
- 135 mg/m2/Week Dose (Phase I Only): All participants in Phase I who received 135 mg/m2/week intravenous NMS-01940153E
- All Treated Participants (Phase I and II; All Dose Levels): Includes all treated participants in the Phase I and Phase II parts of this study, at all dose levels
Arm/Group | 100 mg/m2/Week Dose (Phase I and II) | 135 mg/m2/Week Dose (Phase I Only) | All Treated Participants (Phase I and II; All Dose Levels)
Number analyzed (Participants) | 24 | 6 | 30
events
  Hemoglobin Decreased | 13 | 5 | 18
  Neutrophil Count Decreased | 6 | 4 | 10
  WBC Decreased | 8 | 6 | 14
  Platelet Count Decreased | 6 | 4 | 10

6. Secondary Outcome: Neutrophils Count Decrease: Time to First Occurrence of >=Grade 3 and Time to Recovery to Grade 1
Description: The mean days to first occurrence of neutrophil count decrease are presented for all dose levels.
  Grade 0: ≥2,000/mm3 Grade 1: ≥1,500-< 2,000/mm3 Grade 2: ≥1,000- < 1,500/mm3 Grade 3: ≥500- < 1,000/mm3 Grade 4: <500/mm3
  * G3 = Time (days) to Treatment Start to First Occurrence of Neutrophil Count Decrease >=Grade 3
  * G3 to Recovery to G1 = Time (days) to First Occurrence of Neutrophil Count Decrease >= Grade 3 to Recovery to Grade 1
Time Frame: From screening to 28 days follow-up, an average 6 months
Population: Only participants who experienced G3 or G4 were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 100 mg/m2/Week Dose (Phase I and II) | 135 mg/m2/Week Dose (Phase I Only) | All Treated Participants (Phase I and II; All Dose Levels)
Number analyzed (Participants) | 2 | 4 | 6
days
  >=G3 | 63.00 (19.80) | 28.00 (15.36) | 39.67 (23.38)
  >= G3 to Recovery to G1 | 7.00 (1.41) | 7.33 (3.51) | 7.20 (2.59)

7. Secondary Outcome: Blood Chemistry: Treatment-emergent Abnormalities by Dose Level
Description: Treatment-emergent abnormalities in blood chemistry at any grade are presented by dose level.
  ALP = Alkaline phosphatase ALT = Alanine aminotransferase AST = Aspartate aminotransferase GGT = Gamma-glutamyl transferase LDH = Lactate dehydrogenase
Time Frame: From screening to 28 days follow-up, an average 6 months
Population: All treated participants
Measure: Number; unit: events
Arm/Group | 100 mg/m2/Week Dose (Phase I and II) | 135 mg/m2/Week Dose (Phase I Only) | All Treated Participants (Phase I and II; All Dose Levels)
Number analyzed (Participants) | 24 | 6 | 30
events
  Hypoalbuminemia | 8 | 4 | 12
  Hypoglycemia | 0 | 1 | 1
  AST Increased | 12 | 3 | 15
  ALT Increased | 8 | 2 | 10
  GGT Increased | 9 | 1 | 10
  Creatinine Increased | 6 | 3 | 9
  Blood Bilirubin Increased | 7 | 1 | 8
  ALP Increased | 10 | 1 | 11
  Blood LDH Increased | 14 | 4 | 18
  Hypocalcemia | 1 | 1 | 2
  Hypernatremia | 0 | 1 | 1
  Hyperkalemia | 7 | 0 | 7
  Hypomagnesemia | 5 | 3 | 8

8. Secondary Outcome: Blood Chemistry and Coagulation: Treatment-emergent Abnormalities
Description: Treatment Emergent abnormalities by dose Level are presented for blood chemistry and coagulation parameters.
  INR = international normalized ratio LNL = lower normal limit NL = normal limit ULN = upper limit of normal
Time Frame: From screening to 28 days follow-up, an average 6 months
Population: All treated participants
Measure: Number; unit: events
Arm/Group | 100 mg/m2/Week Dose (Phase I and II) | 135 mg/m2/Week Dose (Phase I Only) | All Treated Participants (Phase I and II; All Dose Levels)
Number analyzed (Participants) | 24 | 6 | 30
events
  Hyponatremia: Total | 4 | 2 | 6
  Hyponatremia: Below LNL | 4 | 2 | 6
  Hypokalemia: Total | 0 | 1 | 1
  Hypokalemia: Below LNL | 0 | 1 | 1
  Phosphatemia: Total | 11 | 2 | 13
  Phosphatemia: Above ULN | 3 | 0 | 3
  Phosphatemia: Below LNL | 7 | 2 | 9
  Phosphatemia: Above/Below NL | 1 | 0 | 1
  Hyperglycemia: Total | 9 | 2 | 11
  Hyperglycemia: Above ULN | 9 | 1 | 10
  Hyperglycemia: Above/Below NL | 0 | 1 | 1
  Blood Urea Nitrogen: Total | 2 | 0 | 2
  Blood Urea Nitrogen: Above ULN | 2 | 0 | 2
  Urea: Total | 6 | 0 | 6
  Urea: Above ULN | 5 | 0 | 5
  Urea: Below LNL | 1 | 0 | 1
  Unconjugated Bilirubin: Total | 3 | 0 | 3
  Unconjugated Bilirubin: Above ULN | 3 | 0 | 3
  Total Protein: Total | 7 | 2 | 9
  Total Protein: Above ULN | 2 | 0 | 2
  Total Protein: Below LNL | 4 | 2 | 6
  Total Protein: Above/Below NL | 1 | 0 | 1
  INR: Total | 11 | 1 | 12
  INR: Above ULN | 8 | 1 | 9
  INR: Below LNL | 1 | 0 | 1
  INR: Above/Below NL | 2 | 0 | 2

9. Secondary Outcome: Electrocardiogram Abnormalities
Description: The number of participants who experienced electrocardiogram abnormalities are presented.
Time Frame: From screening to 28 days follow-up, an average 6 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I) | Phase II (Evaluable Population)
Number analyzed (Participants) | 6 | 6 | 18
Participants | 0 | 0 | 0

10. Secondary Outcome: Tmax and Tlast of NMS-01940153E
Description: Plasma pharmacokinetic (PK) profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  Tmax = Time to maximum observed plasma concentration Tlast = Time of last detectable concentration
Time Frame: Day 1 to Day 15
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: hours
Groups:
- 100 mg/m2/Week Dose (Phase I Only): All participants in Phase I who received 100 mg/m2/week intravenous NMS-01940153E
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
hours
  Tmax: Day 1 | 0.933 (0.0327) | 1.19 (0.513)
  Tmax: Day 15: number analyzed (Participants) | 4 | 6
  Tmax: Day 15 | 1.10 (0.216) | 1.87 (1.90)
  Tlast: Day 1 | 169 (3.01) | 154 (39.2)
  Tlast: Day 15: number analyzed (Participants) | 4 | 6
  Tlast: Day 15 | 144 (48.5) | 169 (0.418)

11. Secondary Outcome: Cmax and Clast of NMS-01940153E
Description: Plasma pharmacokinetic (PK) profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  Cmax = Maximum observed plasma concentration Clast = Last detectable concentration
Time Frame: Day 1 to Day 15
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
μM
  Cmax: Day 1 | 0.754 (0.174) | 1.91 (0.640)
  Cmax: Day 15: number analyzed (Participants) | 4 | 6
  Cmax: Day 15 | 1.35 (1.10) | 1.59 (1.31)
  Clast: Day 1 | 0.0590 (0.0191) | 0.0840 (0.0335)
  Clast: Day 15: number analyzed (Participants) | 4 | 6
  Clast: Day 15 | 0.113 (0.0454) | 0.133 (0.0779)

12. Secondary Outcome: AUClast, AUCweekly, and AUCinf of NMS-01940153E
Description: Plasma pharmacokinetic (PK) profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion. Infusions occurred on Days 1, 8, and 15.
  AUClast = Area under the interpolated observed plasma time-concentration curve from infusion start to the last observed plasma concentration AUCweekly = Area under the interpolated observed plasma time-concentration curve from infusion start to 168 hours AUCinf = Area under the interpolated observed plasma time-concentration curve from infusion start extrapolated to infinity based on the last observed plasma concentration
Time Frame: From Days 1 to 21 (168 hours after the Day 15 infusion)
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: h·μM
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
h·μM
  AUClast: Day 1 | 20.8 (4.31) | 24.8 (8.55)
  AUClast: Day 15: number analyzed (Participants) | 4 | 6
  AUClast: Day 15 | 30.0 (9.16) | 39.1 (14.9)
  AUCweekly: Day 1 | 20.8 (4.35) | 25.7 (7.11)
  AUCweekly: Day 15: number analyzed (Participants) | 4 | 6
  AUCweekly: Day 15 | 32.4 (6.49) | 39.0 (14.8)
  AUCinf: Day 1 | 28.7 (6.88) | 37.1 (14.9)
  AUCinf: Day 15: number analyzed (Participants) | 4 | 6
  AUCinf: Day 15 | 48.1 (19.6) | 62.9 (34.1)

13. Secondary Outcome: t½,z of NMS-01940153E
Description: Plasma pharmacokinetic (PK) profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  t½,z = Half-life of the terminal phase of observed plasma concentration
Time Frame: Day 1 to Day 15
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
days
  t½,z Day 1 | 3.74 (0.800) | 4.17 (1.40)
  t½,z Day 15: number analyzed (Participants) | 4 | 6
  t½,z Day 15 | 4.38 (2.64) | 4.79 (1.15)

14. Secondary Outcome: CL and CLss of NMS-01940153E
Description: Plasma pharmacokinetic (PK) profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  CL = Clearance based on last observed concentration and extrapolation to infinity CLss = Clearance calculated for a dosing period of 168 h either after a single dose or in steady-state
Time Frame: Day 1 to Day 15
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
L/h
  CL: Day 1 | 10.1 (3.16) | 10.2 (4.01)
  CL: Day 15: number analyzed (Participants) | 4 | 6
  CL: Day 15 | 6.12 (2.24) | 6.19 (2.08)
  CLss: Day 1 | 13.8 (4.14) | 13.8 (3.73)
  CLss: Day 15: number analyzed (Participants) | 4 | 6
  CLss: Day 15 | 8.53 (2.50) | 9.31 (2.52)

15. Secondary Outcome: Vss and Vss,SS of NMS-01940153E
Description: Plasma pharmacokinetic (PK) PK profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  Vss = Volume of distribution at steady state based last observed concentration extrapolated to infinity and Clearance calculated for a dosing period of 168 h either after a single dose or in steady-state Vss,SS = Volume of distribution at steady state based last observed concentration extrapolated to infinity and clearance based on last observed concentration and extrapolation to infinity
Time Frame: Day 1 to Day 15
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
L
  Vss: Day 1 | 1230 (395) | 1210 (199)
  Vss: Day 15: number analyzed (Participants) | 4 | 6
  Vss: Day 15 | 787 (304) | 919 (245)
  Vss,SS: Day 1 | 1700 (620) | 1630 (285)
  Vss,SS: Day 15: number analyzed (Participants) | 4 | 6
  Vss,SS: Day 15 | 1180 (649) | 1380 (354)

16. Secondary Outcome: RA AUCweekly and RA Cmax of NMS-01940153E
Description: Plasma pharmacokinetic (PK) PK profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion. Infusions occurred on Days 1, 8, and 15.
  RA AUCweekly = Accumulation ratio Day 1 to 15 calculated using area under the interpolated observed plasma time-concentration curve from infusion start to 168 hours RA Cmax = Accumulation ratio Day 1 to 15 calculated using maximum observed plasma concentration
Time Frame: Day 21 (168 hours after the Day 15 infusion)
Population: All Phase I participants
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
ratio
  RA AUCweekly: Day 15: number analyzed (Participants) | 4 | 6
  RA AUCweekly: Day 15 | 1.66 (0.188) | 1.51 (0.293)
  RA Cmax: Day 15: number analyzed (Participants) | 4 | 6
  RA Cmax: Day 15 | 1.78 (1.36) | 0.858 (0.547)

17. Secondary Outcome: FE of NMS-01940153E
Description: Urine pharmacokinetic profiles of NMS-01940153E were characterized on Day 1 and 15 of the first Cycle after infusion.
  FE = Molar fraction of excreted compound relative to the administered molar dose calculated using urine concentration and volume data
Time Frame: Day 1 to Day 15
Population: All treated participants
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 100 mg/m2/Week Dose (Phase I Only) | 135 mg/m2/Week Dose (Phase I Only)
Number analyzed (Participants) | 6 | 6
percentage
  FE Day 1 | 0.458 (0.374) | 0.357 (0.260)
  FE Day 15: number analyzed (Participants) | 4 | 6
  FE Day 15 | 0.563 (0.424) | 0.826 (0.713)

18. Secondary Outcome: Phase I Objective Tumor Response (Partial and Complete Response)
Description: Phase I any dose level, objective response and best overall tumor response are presented, as measured by investigator assessed RECIST 1.1 (Phase I).
  The objective response rate was calculated as the proportion of evaluable patients who achieved best overall response (BOR), confirmed complete response (CR) or partial response (PR).
Time Frame: Phase I: From the Study Start Date to Phase I Completion (32 months)
Population: Treated Patients with at Least One RECIST 1.1 On-Treatment Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I)
Number analyzed (Participants) | 6 | 5
Participants
  Objective Response (Partial Response) | 1 | 1
  Objective Response (Complete Response) | 0 | 0
  Stable Disease | 1 | 2
  Progressive Disease | 4 | 2

19. Secondary Outcome: Phase II Objective Response Rate as Measured by Investigator-assessed mRECIST
Description: Objective response rate as measured by investigator-assessed mRECIST in Phase II.
Time Frame: Phase II: From Phase II start to Study Completion (23 months)
Population: Evaluable participants with at least one mRECIST Assessment on Treatment were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Treated Participants: All participants in Phase II who received 100 mg/m2/week intravenous NMS-01940153E and with at least one mRECIST Assessment on Treatment
Arm/Group | Phase II Treated Participants
Number analyzed (Participants) | 14
Participants
  Stable Disease | 3
  Progressive Disease | 11
  Objective Response (Partial Response) | 0
  Objective Response (Complete Response) | 0

20. Secondary Outcome: Phase I: Duration of Response (DoR) as Measured by Investigator-assessed RECIST 1.1
Description: Duration of response (DoR) as measured by investigator-assessed Response evaluation criteria in solid tumours (RECIST) 1.1.
  Duration of Response (months): was time in months from response start date to either date of disease progression/death due to progression of disease. It was calculated only for participants with complete response or partial response as best overall response.
Time Frame: Phase I: From the Study Start Date to Phase I Completion (32 months)
Population: Phase I participants who experienced partial response
Measure: Number; unit: months
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I)
Number analyzed (Participants) | 1 | 1
months | 2.6 | 9.3

21. Secondary Outcome: Phase II: Duration of Response (DoR) as Measured by Investigator-assessed RECIST 1.1. and Investigator-assessed mRECIST
Description: Duration of response (DoR) as measured by investigator-assessed Response evaluation criteria in solid tumours (RECIST) 1.1 and investigator-assessed modified RECIST (mRECIST).
  Duration of Response (months): was time in months from response start date to either date of disease progression/death due to progression of disease. It was calculated only for participants with complete response or partial response as best overall response.
Time Frame: Phase II: From Phase II start to Study Completion (23 months)
Population: Phase II Evaluable Population. No participants had a RECIST or mRECIST complete or partial response observed.
Arm/Group | Phase II (Evaluable Population)
Number analyzed (Participants) | 0

22. Secondary Outcome: Progression Free Survival, as Measured by Investigator-assessed RECIST 1.1, in Phases I and II
Description: Progression Free Survival as measured by investigator assessed RECIST 1.1, for all treated participants in Phase I and Phase II.
  Phase 2 started before Phase 1 completed.
Time Frame: as for outcome 3
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I) | Phase II (Evaluable Population)
Number analyzed (Participants) | 6 | 6 | 14
months | 1.9 [1.7 to 6.5] | 7.8 [1.8 to 25.1] | 1.9 [1.8 to 4.1]

23. Secondary Outcome: Overall Survival in Phases I and II
Description: Overall Survival for all treated participants in Phases I and II. The estimates are based on the Kaplan-Meier (KM) method.
  Phase 2 started before Phase 1 completed.
Time Frame: as for outcome 3
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg/m2/Week Dose (Phase I) | 135 mg/m2/Week Dose (Phase I) | Phase II (Evaluable Population)
Number analyzed (Participants) | 6 | 6 | 14
months | 9.7 [5.2 to NA] — Insufficient number of participants with events | 15.7 [4.7 to NA] — Insufficient number of participants with events | 7.3 [3.9 to NA] — Insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Phase I: From the Study Start Date to Phase I Completion (32 months) - Phase II: From Phase II start to Study Completion (23 months). Phase 2 started before Phase 1 completed.
Description: Adverse events were coded by MedDRA and severity was graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
  For non-serious AEs, the number of participants who experienced at least 1 occurrence of a treatment-emergent non-serious AEs, by MedDRA System Organ Class and Preferred Term are presented.
  The one participant who was enrolled but not treated was not assessed for adverse events and therefore this cohort has not been included.
Groups:
- Phase I: 100 mg/m2/Week: All participants in Phase I who received 100 mg/m2/week intravenous NMS-01940153E
- Phase I: 135 mg/m2/Week: All participants in Phase I who received 135 mg/m2/week intravenous NMS-01940153E
- Phase II: 100 mg/m2/Week: All participants in Phase II who received 100 mg/m2/week intravenous NMS-01940153E
Arm/Group | Phase I: 100 mg/m2/Week | Phase I: 135 mg/m2/Week | Phase II: 100 mg/m2/Week
All-Cause Mortality (participants affected / at risk) | 5/6 | 5/6 | 9/18
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 5/18
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 100 mg/m2/Week (N=6) | Phase I: 135 mg/m2/Week (N=6) | Phase II: 100 mg/m2/Week (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 100 mg/m2/Week (N=6) | Phase I: 135 mg/m2/Week (N=6) | Phase II: 100 mg/m2/Week (N=18)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (8)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3)
Asthenia (General disorders) | 1 (2) | 1 (1) | 8 (10)
Infusion site reaction (General disorders) | 1 (1) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 3 (6) | 2 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (7) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (12) | 2 (2) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (15)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Burn infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
In the Phase II part of the study, among the patients evaluable for efficacy, no objective response (partial response or clinical response) was observed at the first futility analysis. Therefore, this study was terminated for clinical futility, according to the protocol rules.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT05630937/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05630937/SAP_003.pdf